CLINICAL TRIAL: NCT02732886
Title: A Pilot Study to Compare Efficacy of Medifoam® and Betafoam® as a New Dressing Including Povidone-iodine, in Patients With Diabetes Foot Ulcer
Brief Title: Betafoam Diabetes Mellitus Foot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mundipharma Korea Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTF15-KR-402
Record Dates: First submitted 2016-03-15; First posted 2016-04-11 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Diabetes Mellitus; Foot Ulcer
Keywords: foam dressing
MeSH Terms: conditions — Diabetes Mellitus; Foot Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Betafoam® (Experimental): Brand name: Betafoam® Generic term: Wound dressing with 3% povidone iodine
  Interventions: Device: Betafoam®
- Medifoam® (Active Comparator): Brand name: Medifoam® Generic term: Wound dressing
  Interventions: Device: Medifoam®

INTERVENTIONS:
Device: Medifoam® — Foam Dressing
  Other Names: Medifoam
  Arms: Medifoam®
Device: Betafoam® — Foam dressing including Betadine iodine
  Other Names: Betafoam
  Arms: Betafoam®

SUMMARY:
This study is to compare the efficacy and safety of Medifoam® and Betafoam®, which is a new dressing that contains povidone-iodine, in patients with diabetes foot ulcer. 70 patients (35 each arm) are targeted to be enrolled in this study. Treatment follow periods are 8weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult of age ≥19 years at the time of informed consent
* Foot ulcers related to diabetes mellitus:

  * Present
  * Type I or II diabetes mellitus with HbA1c <10%, or serum creatinine ≤ 200 μmol/l
  * Wagner grade I-II (Partial- or full- thickness and not involving bone, tendon, or capsule (probing to tendon or capsule)
  * Post -debridement ulcer bed size ≥ 1*1cm2
* No clinical signs of infection & necrosis
* Site at anywhere below ankle
* No vascular abnormalities of the foot by palpation (i.e. the dorsalis pedis should be examined by the physician and characterized as present or absent)

Exclusion Criteria:

* Pregnant & lactating females
* Known allergy to the dressing product including povidone iodine
* Known hyperthyroidism or other acute thyroid diseases
* Subject with clinical infection who should be administered antibiotics continuously after enrolment
* Subject has any condition(s) that seriously compromises the patient's ability to complete this study.
* Subject has participated in interventional study utilizing an investigational drug within the previous 30 days
* Subjects with known immune-suppressed state; who undergo chemotherapy or with end-stage renal disease requiring haemodialysis or had kidney transplant surgery previously and with immunosuppressant specifically
* Subjects requiring skin grafting per physician's discretion
* Vulnerable subjects as defined by Good Clinical Practice guidelines.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2016-03-29 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with a target ulcer which achieves complete wound closure in 8 weeks | 8 weeks
  Skin re-epithelialization without drainage or dressing requirements

SECONDARY OUTCOMES:
Proportion of subjects with a target ulcer which achieves complete wound closure in 4 weeks | 4 weeks
  Skin re-epithelialization without drainage or dressing requirements
Wound infection rate until completion of skin re-epithelialization | 8 weeks
  Wound infection rate until the completion of skin re-epithelialization in each subject by recording the signs and symptoms of infection at every visit
Patient's level of satisfaction with treatment measured weekly using numeric rating scale (NRS) | 8 weeks
  Level of patient's satisfaction with the application and removal of dressing, as measured using numeric rating scale (NRS). This is done weekly from Visits 3 to 17.
Number of days till completion of wound healing from baseline | 8 weeks
Total number of the dressing change and mean number of dressing change per day compared to wound healing period | 8 weeks
Safety as determined through collection of adverse events | 8 weeks
Change amount and change rate of the target ulcer size after using the investigational device | 8 weeks
  The area of the target ulcer is calculated with a film drawn to the shape of the wound at the target ulcer, by using the Visitrak digital planimetry.

CONTACTS AND LOCATIONS:
Overall Officials: Hyongjin Jung, Dr. PhD., Principal Investigator — Inje University Sangye Paik Hospital,
Locations (1):
- Inje University Sanggye Paik Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gwak HC, Han SH, Lee J, Park S, Sung KS, Kim HJ, Chun D, Lee K, Ahn JH, Kwak K, Chung HJ. Efficacy of a povidone-iodine foam dressing (Betafoam) on diabetic foot ulcer. Int Wound J. 2020 Feb;17(1):91-99. doi: 10.1111/iwj.13236. Epub 2019 Nov 26. PMID 31773882